CLINICAL TRIAL: NCT03065855
Title: Amonocenter, Prospective, Randomized Clinical Trial to Investigate the Removal Time of Urinary Catheter After Laparoscopic Anterior Resection of the Rectum.
Brief Title: Removal Time of Urinary Catheter After Laparoscopic Anterior Resection of the Rectum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARCTIC
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Rectum Cancer
Keywords: laparoscopic mesorectal excision; rectal cancer; urinary distention
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early removal group (Experimental): All participants are to have a urethral catheter placed following successful placement of an epidural catheter for analgesia prior. Following urethral catheter placement participants will be randomly assigned to either the experimental arm or the control arm. Participants assigned to the experimental arm will have their urethral catheters removed at 2 days following surgery.
  Interventions: Procedure: Early removal group
- Normal removal group (Active Comparator): All participants are to have a urethral catheter placed following successful placement of an epidural catheter for analgesia prior. Following urethral catheter placement participants will be randomly assigned to either the experimental arm or the control arm. Participants assigned to the control group will have their urethral catheters removed at 7days following surgery, as is standard practice in our institution.
  Interventions: Procedure: Normal removal group

INTERVENTIONS:
Procedure: Early removal group — Participants assigned to the experimental arm will have their urethral catheters removed at 2 days after after laparoscopic anterior resection of the rectum.
  Arms: Early removal group
Procedure: Normal removal group — Participants assigned to the control group will have their urethral catheters removed at 7days following surgery, as is standard practice in our institution.
  Arms: Normal removal group

SUMMARY:
Traditionally these catheters are retained for 7 days, because a higher incidence of urinary retention is related to early removal of the urinary catheter. However, recently Enhanced Recovery After Surgery presents that urinary catheters placed via the urethra can be withdrawn 48 hours after colon/rectal surgery in patients receiving epidural pain relief，but there is no clear data on the incidence of urine retention.Longer retaining time of urethral catheter would induce the urinary tract infection while early removal of urethral catheter is considered to develop acute retention of urine due to lack of sensation when the bladder is full. Taking the comfort and mobility for faster rehabilitation of patients into account, the investigators aim at obtain the optimal removal time of urinary catheter after after laparoscopic anterior resection of the rectum

DETAILED DESCRIPTION:
For a better view to avoid accidental trauma and monitoring kidney function during surgery and in the post-surgery period, patients undergoing abdominal operations will usually have a urinary catheter placed in the bladder before the surgery. Traditionally these catheters are retained for 7 days, because a higher incidence of urinary retention is related to early removal of the urinary catheter. However, recently Enhanced Recovery After Surgery presents that urinary catheters placed via the urethra can be withdrawn 48 hours after colon/rectal surgery in patients receiving epidural pain relief.

Longer retaining time of urethral catheter would induce the urinary tract infection while early removal of urethral catheter is considered to develop acute retention of urine due to lack of sensation when the bladder is full. Taking the comfort and mobility for faster rehabilitation of patients into account, the investigators aim at obtain the optimal removal time of urinary catheter after after laparoscopic anterior resection of the rectum

.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to consent to participate in trial
2. Patients with rectal cancer who underwent total or tumor-specific-mesorectal excision with colorectal or colonanal anastomosis
3. Elective surgery
4. ASA classification of 1~3
5. If male, international prostate symptom score <20.

Exclusion Criteria:

1. Combined pelvic surgery(pelvic lymph node dissection, hysterectomy, salpingo-oophorectomy, posterior vaginectomy, cystectomy, ureteral double-J stenting, ureterectomy, ureteroureterostomy, prostatectomy)
2. Postoperative complications with a Dindo grade III or more
3. Known urinary disease(end-stage renal disease, benign prostatic hyperplasia, neurogenic bladder, malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Post-operative urinary retention requiring re-catheterisation | 1 day following urethral catheter removal
  Development of acute post-operative urinary retention demonstrated by a post-void residual >100mls on bladder ultrasound requiring re-catheterisation within 1 day of removal of urethral catheter in the post-operative period

SECONDARY OUTCOMES:
Urinary tract infection | Within 7 days of urethral catheter removal
  Before catheter removal, take a mid-stream urine sample for microscopy and culture. Leucocyte in urine ≥5/HP for man and ≥10/HP for woman is defined as bacteruria with urinary irritation or not.A pure culture of a single organism of >100,000 colony forming units will be considered a positive culture.
Urethrorrhagia | Within 7 days of urethral catheter removal
  take a mid-stream urine sample for Clinical urine tests and RBC≥3/HP is defined as urethrorrhagia.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Other researchers have access to data in the form of published papers

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246
- [Derived] Xu L, Tao ZY, Lu JY, Zhang GN, Qiu HZ, Wu B, Lin GL, Xu T, Xiao Y. A single-center, prospective, randomized clinical trial to investigate the optimal removal time of the urinary catheter after laparoscopic anterior resection of the rectum: study protocol for a randomized controlled trial. Trials. 2019 Feb 15;20(1):133. doi: 10.1186/s13063-019-3210-1. PMID 30770766